CLINICAL TRIAL: NCT02893735
Title: A Prospective 4-year Clinical Study Evaluating Two Resin Composites on Diastema Closure and Reshaping
Brief Title: Clinical Comparison of Two Resin Composites on Diastema Closure and Reshaping at Four Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zeynep Bilge Kutuk, PhD, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014/03-4(KA-14004)
Record Dates: First submitted 2016-08-05; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Diastema
Keywords: Clinical Trial; Composite resin
MeSH Terms: conditions — Diastema | interventions — Filtek Z550

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Charisma-Diamond (Active Comparator): Charisma Diamond was randomly applied for diastema closure.
  Interventions: Other: Charisma-Diamond
- Filtek-Z550 (Active Comparator): Filtek-Z550 was randomly applied for diastema closure.
  Interventions: Other: Filtek-Z550

INTERVENTIONS:
Other: Charisma-Diamond — The surfaces were etched using 35% phosphoric acid for 30 s. The etched surfaces were rinsed and dried. Nano-hybrid resin composite system was used Charisma-Diamond in combination Gluma2 Bond etch&rinse adhesive. The composite increments were carefully placed between the matrix strip and tooth by using a hand instrument. The composite resin restorations were light-cured (600 mW/cm²). Occlusion was checked with thin articulating papers. Restoration surfaces were finished and polished with fine finishing diamond burs, stones and rubber cups whereas; proximal and labial surfaces were contoured and polished with finishing strips. The treatments were completed by instructing the patients about the oral hygiene measures for cleaning their restorations with toothbrush and dental floss.
  Arms: Charisma-Diamond
Other: Filtek-Z550 — The surfaces were etched using 35% phosphoric acid for 30 s. The etched surfaces were rinsed and dried. Nano-hybrid resin composite system was used Filtek-Z550 in combination with Adper™ Single Bond 2 etch&rinse adhesive. The composite increments were carefully placed between the matrix strip and tooth by using a hand instrument. The composite resin restorations were light-cured (600 mW/cm²). Occlusion was checked with thin articulating papers. Restoration surfaces were finished and polished with fine finishing diamond burs, stones and rubber cups whereas; proximal and labial surfaces were contoured and polished with finishing strips. The treatments were completed by instructing the patients about the oral hygiene measures for cleaning their restorations with toothbrush and dental floss.
  Arms: Filtek-Z550

SUMMARY:
The aim of this study was to evaluate the clinical performances of nano-hybrid resin composite systems used for anterior diastema closure and tooth reshaping at 4 years in service using FDI Criteria.

Twenty-three patients with diastema problem were enrolled. Nano-hybrid resin composites to be used on each patient were randomly selected. Thirty-seven teeth (10 patients) were restored with Filtek-Z550 (3M/ESPE) in combination with Adper™ Single Bond 2 (3M/ESPE) in Group 1; whereas 39 teeth (13 patients) were restored with Charisma-Diamond (Heraeus Kulzer) in combination with Gluma2 Bond (Heraeus Kulzer) in Group 2, by two operators. Esthetic, functional and biological properties of the restorations were evaluated at baseline, 1-4 years using FDI Criteria establishing a score-range of 1-5. The data were evaluated using the Fisher's Chi-Square (p=0.05).

DETAILED DESCRIPTION:
The aim of this study was to evaluate the clinical performances of nano-hybrid resin composite systems used for anterior diastema closure and tooth reshaping at 4 years in service using FDI Criteria.

The study protocol was approved by the Ethical Committee of Hacettepe University, Ankara, Turkey and the Ethical Committee of Ministry of Health (protocol HEK KA-14004). A total of 23 patients (6 male, 17 female, mean age: 31.27) with maxillary anterior midline or multi-diastema problem received 76 direct composite resin restorations.

The teeth to be restored were first cleaned with pumice-water slurry using a rubber cup. The appropriate shade of restorative material was selected using a standard VITAPAN® Classic shade guide and initial intraoral photographs were taken. Teeth were then isolated using cotton rolls and Mylar strips were placed with the help of wedges interproximally to achieve a smooth and overhang free restoration outline in the cervical area and to form final restorations. The surfaces to be restored were etched using 35% phosphoric or orthophosphoric acid for 30 s according to the restorative system used. The etched surfaces were rinsed and dried. Nano-hybrid resin composite systems to be used on each patient were randomly selected. Thirty seven teeth of 10 patients were restored with Filtek-Z550 (3M/ESPE, St. Paul, MN, USA) in combination with Adper™ Single Bond 2 (3M/ESPE, St. Paul, MN, USA) etch&rinse adhesive; whereas 39 teeth of 13 patients were restored with Charisma-Diamond (Heraeus Kulzer, GmbH, Germany) in combination with Gluma2 Bond (Heraeus Kulzer, GmbH, Germany) etch&rinse adhesive by two operators. Materials were used according to the manufacturers' instructions. Two calibrated observers who were blinded to the objective of this study performed the evaluations. For maximum validity, the observers were calibrated by using the web-based training and calibration tool www.e-calib.info recommended by FDI. Both observers evaluated the esthetic, functional and biological properties of the restorations independently at baseline, 1-2-3 and 4 years using FDI Criteria establishing a score-range of 1-5 (1-Clinically excellent/very good, 2-Clinically good, 3-Clinically sufficient/satisfactory, 4-Clinically unsatisfactory and 5-Clinically poor). After data collection, in case of discrepancies in scoring, restorations were evaluated again, a consensus was reached and this was accepted as the final score.

Statistical analysis was performed with SPSS 15.0 software. To compare the performance of restorative materials according to FDI criteria over the study period, the Fisher's Chi-Square test was used. The Cochran's Q test was then used to compare the 1-2-3 and 4-year scores of each material with baseline scores to evaluate the changes of each dependent group by the time. Survival curves were obtained using Kaplan-Meier method. p values less than 0.05 were considered to be statistically significant in all tests.

ELIGIBILITY:
Inclusion Criteria:

* all subjects were required to be at least 18 years old,
* able to read and sign the informed consent document,
* physically and psychologically able to tolerate conventional restorative procedures,
* having no active periodontal or pulpal diseases,
* having teeth with good restorations, and
* willing to return for follow-up examinations as outlined by the investigators.

Exclusion Criteria:

* uncontrolled parafunction;
* insufficient oral hygiene leading to caries lesions more than twice yearly during the previous 2 years;
* being pregnant or nursing; and
* having periodontal or gingival disease.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2011-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Clinical performance of restorations, graded on a 5-point scale, using FDI criteria | Change from baseline to 4 year outcome of restorations were evaluated.
  This outcome may be classified as "1-Clinically excellent/ very good", "2-Clinically good (after correction, very good)", "3-Clinically sufficient/ satisfactory (minor shortcomings with no adverse effects but not adjustable without damage to the tooth)", "4-Clinically unsatisfactory (repair for prophylactic reasons)", "5-Clinically poor (replacement necessary)" classification of the Esthetic, Functional and Biological properties

SECONDARY OUTCOMES:
Surface Luster, graded on a 5-point scale (FDI criteria) | Change from baseline to 4 year outcome of restorations were evaluated.
  May be classified as "Luster comparable to enamel", "Slightly dull, not noticeable from speaking distance", "Dull surface but acceptable if covered with film of saliva", "Rough surface, cannot be masked by saliva film, simple polishing is not sufficient. Further intervention necessary", "Quite rough, unacceptable plaque retentive surface"
Staining margin, graded on a 5-point scale (FDI criteria) | Change from baseline to 4 year outcome of restorations were evaluated.
  May be classified as "No surface staining", "Minor staining, easily removable", "Moderate surface staining, also present on other teeth, not aesthetically unacceptable", "Surface staining present on the restoration and is unacceptable; major intervention necessary for improvement", "Severe staining and/or subsurface staining (generalized or localized); not accessible for intervention"
Colour stability and translucency, graded on a 5-point scale (FDI criteria) | Change from baseline to 4 year outcome of restorations were evaluated.
  May be classified as "Good colour match no difference in shade and translucency", "Minor deviations", "Clear deviation but acceptable. Does not affect aesthetics", "(Localised) clinically unsatisfactory but can be corrected by repair", "Unacceptable. Replacement necessary"
Fractures and Retention, graded on a 5-point scale (FDI criteria) | Change from baseline to 4 year outcome of restorations were evaluated.
  May be classified as "Restoration retained, no fractures/cracks", "Small hairline crack", "Two or more or larger hairline cracks and/or chipping(not affecting the marginal integrity or proximal contact", "Chipping fractures which damage marginal quality or proximal contacts; bulk fractures with or without partial loss(less than half of the restoration)", "Partial or complete loss of restoration"
Marginal Adaptation, graded on a 5-point scale (FDI criteria) | Change from baseline to 4 year outcome of restorations were evaluated.
  May be classified as "Harmonious outline, no gaps, no discoloration", "Marginal gap (50 µm) or Small marginal fracture removable by polishing", "Gap< 150 µm not removable or Severe small enamel or dentin fractures", "Gap> 250 µm or dentine exposed or Chip fracture damaging margins or Notable enamel or dentine wall fracture", "Filling is loose but in situ"
Postoperative Hypersensibility, tooth vitality, graded on a 5-point scale (FDI criteria) | Change from baseline to 4 year outcome of restorations were evaluated.
  May be classified as "No hypersensitivity, normal vitality", "Low hypersensitivity for a limited period of time, normal vitality", "Premature/slightly more intense or Delayed/weak sensitivity; no subjective complaints, no treatment needed", "Premature/very intense or Extremely delayed/weak with subjective complaints or Negative sensitivity intervention necessary but not replacement", "Very intense, acute pulpitis or no vital. Endodontic treatment is necessary and restoration has to be replaced"
Recurrence of Caries, erosion, abfraction, graded on a 5-point scale (FDI criteria) | Change from baseline to 4 year outcome of restorations were evaluated.
  May be classified as "No secondary or primary caries", "Very small and localized. No operative treatment required", "Larger areas of: Demineralisation or Erosion or Abrasion/abfraction in dentine. Localized and accessible and can be repaired", "Caries with cavitation or Erosion in dentine or Abrasion/abfraction in dentine Localized and accessible and can be repaired", "Deep secondary caries or exposed dentine that is not accessible for repair of restoration"
Tooth integrity (enamel cracks), graded on a 5-point scale (FDI criteria) | Change from baseline to 4 year outcome of restorations were evaluated.
  May be classified as "Complete integrity", "Small margin enamel(<150 µm) or Hairline crack in enamel (<150 µm not probable)", "Enamel split(<250 µm) or Crack< 250 µm, no adverse effects", "Major enamel split (gap>250 µm or dentine or base exposed) or Crack>250 µm (probe penetrates)", "Cusp or tooth fracture"

CONTACTS AND LOCATIONS:
Overall Officials: Sevil Gurgan, PhD, DDS, Study Director — Hacettepe University School of Dentistry
Locations (1):
- Hacettepe University School of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Ergin E, Kutuk ZB, Oztas SS, Cakir FY, Gurgan S. 6-Months Clinical Comparison of Two Resin Composites on Diastema Closure. J Dent Res (Spec Iss 94 A): 599, 2015